CLINICAL TRIAL: NCT05277051
Title: A Phase 1 First-Time-in-Human, Open-Label Study of GSK4381562 Administered as Monotherapy and in Combination With Anticancer Agents in Participants With Selected Advanced Solid Tumors
Brief Title: First-Time-in-Human Study of GSK4381562 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 217228; 2023-509414-11-00 (EU CTIS Number)
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms
Keywords: Advanced solid tumors; Metastatic solid tumor; Anticancer agents; Dostarlimab; Remzistotug; GSK4428859A; Belrestotug; Nelistotug; GSK5764227; Head and neck squamous cell carcinoma (HNSCC); Non-small-cell lung cancer (NSCLC); Breast cancer (BC); Clear cell renal cell cancer (ccRCC); Gastric cancer (GC); Colorectal cancer (CRC); Endometrial cancer (EC); Epithelial ovarian; fallopian tube; and primary peritoneal cancers
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Carcinoma, Renal Cell; Stomach Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Intervention Model Description: 4 Dose Escalation arms (Arm A: remzistotug alone; Arm B: remzistotug plus dostarlimab; Arm C: remzistotug plus dostarlimab plus belrestotug); Arm I: GSK5764227 plus dostarlimab) and 5 other arms, Arm D (dostarlimab plus belrestotug; Arm E (dostarlimab plus belrestotug plus remzistotug Arm F (dostarlimab plus belrestotug plus nelistotug; Arm G (China cohort: dostarlimab);
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Participants Receiving remzistotug Monotherapy (Arm A) (Experimental)
  Interventions: Drug: Remzistotug
- Participants Receiving remzistotug Plus Dostarlimab (Arm B) (Experimental)
  Interventions: Drug: Remzistotug; Drug: Dostarlimab
- Participants Receiving remzistotug Plus Dostarlimab Plus belrestotug (Arm C) (Experimental)
  Interventions: Drug: Remzistotug; Drug: Dostarlimab; Drug: Belrestotug
- Participants Receiving Dostarlimab Plus belrestotug (Arm D) (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Belrestotug
- Participants Receiving dostarlimab Plus belrestotug Plus remzistotug (Arm E) (Experimental)
  Interventions: Drug: Remzistotug; Drug: Dostarlimab; Drug: Belrestotug
- Participants Receiving dostarlimab Plus belrestotug Plus nelistotug (Arm F) (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Belrestotug; Drug: Nelistotug
- China Cohort: Participants receiving dostarlimab (Arm G) (Experimental)
  Interventions: Drug: Dostarlimab
- Participants Receiving GSK5764227 Plus dostarlimab (Arm I) (Experimental)
  Interventions: Drug: Dostarlimab; Drug: GSK5764227

INTERVENTIONS:
Drug: Remzistotug — Remzistotug will be administered.
  Arms: Participants Receiving dostarlimab Plus belrestotug Plus remzistotug (Arm E); Participants Receiving remzistotug Monotherapy (Arm A); Participants Receiving remzistotug Plus Dostarlimab (Arm B); Participants Receiving remzistotug Plus Dostarlimab Plus belrestotug (Arm C)
Drug: Dostarlimab — Dostarlimab will be administered.
  Arms: China Cohort: Participants receiving dostarlimab (Arm G); Participants Receiving Dostarlimab Plus belrestotug (Arm D); Participants Receiving GSK5764227 Plus dostarlimab (Arm I); Participants Receiving dostarlimab Plus belrestotug Plus nelistotug (Arm F); Participants Receiving dostarlimab Plus belrestotug Plus remzistotug (Arm E); Participants Receiving remzistotug Plus Dostarlimab (Arm B); Participants Receiving remzistotug Plus Dostarlimab Plus belrestotug (Arm C)
Drug: Belrestotug — Belrestotug will be administered.
  Arms: Participants Receiving Dostarlimab Plus belrestotug (Arm D); Participants Receiving dostarlimab Plus belrestotug Plus nelistotug (Arm F); Participants Receiving dostarlimab Plus belrestotug Plus remzistotug (Arm E); Participants Receiving remzistotug Plus Dostarlimab Plus belrestotug (Arm C)
Drug: Nelistotug — Nelistotug will be administered.
  Arms: Participants Receiving dostarlimab Plus belrestotug Plus nelistotug (Arm F)
Drug: GSK5764227 — GSK5764227 will be administered.
  Arms: Participants Receiving GSK5764227 Plus dostarlimab (Arm I)

SUMMARY:
This is a first time in-human (FTIH) study designed to investigate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of remzistotug in participants with select loco-regionally recurrent solid tumors or metastatic solid tumors where curative or standard treatment options have been exhausted.

ELIGIBILITY:
Inclusion criteria:

* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) or
  * Is a WOCBP and using a contraceptive method that is highly effective with a failure rate of less than (<)1 percent ([%] per year), during the intervention period and for specified time after end of study treatment.
  * A WOCBP must have a negative highly sensitive pregnancy test within 24-48 hours before the first dose of study intervention.
  * Requirement for Arm I only: Male participants agree to use contraception and for their female partner to use contraception, if applicable.
* Histological or cytological documentation of loco-regionally recurrent solid tumors where curative treatment options have been exhausted, or metastatic solid tumors; types as follows:

  * head and neck squamous cell carcinoma (HNSCC)
  * non-small-cell lung cancer (NSCLC)
  * breast cancer (BC)
  * clear cell renal cell cancer (ccRCC)
  * gastric cancer (GC)
  * colorectal cancer (CRC)
  * endometrial cancer (EC)
  * epithelial ovarian, fallopian tube, and primary peritoneal cancers- Disease that has progressed after standard therapy for the specific tumor type, or for which standard therapy has proven to be ineffective, intolerable, or is considered inappropriate, or if no further standard therapy exists.
  * Measurable disease per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Life expectancy of at least 12 weeks.
* Adequate organ function, as defined in the protocol.
* For participants enrolled in a PK/PD cohort, participant agrees to a fresh tumor biopsy during Screening and at approximately 6-weeks after treatment initiation.

Exclusion Criteria:

* Prior treatment with the following therapies (specified time periods are from last dose of prior treatment to first dose of study intervention):

  * Any therapy directed against Polio virus receptor (PVR)-related immunoglobulin domain-containing (PVRIG) (COM701 or other anti-PVRIG monoclonal antibody [mAb]) or other cluster of differentiation (CD)226 axis receptor (T-cell immunoglobulin and immunoreceptor tyrosine-based inhibition motif domain [TIGIT] or CD96) at any time.
  * For Arm I only, prior treatment with orlotamab, enoblituzumab, I-Dxd, or other B7-H3 targeted agents.
  * Other prior immunotherapy, chemotherapy, targeted therapy, biological therapy or radiation therapy within specified periods as defined in the protocol.
  * Investigational therapy: if the participant has participated in a clinical study and has received an investigational product within 4 weeks or 5 half-lives of the investigational product (whichever is shorter).
* Prior allogenic or autologous bone marrow transplantation or other solid organ transplantation.
* Toxicity from previous anticancer treatment, including:

  * Greater than or equal to Grade 3 immune-mediated toxicity considered related to prior immunotherapy and that led to treatment discontinuation; or
  * History of myocarditis of any grade during a previous treatment with immunotherapy
  * Toxicity related to prior treatment that has not resolved to less than or equal to (<=) Grade 1. Non clinically relevant Grade 2 toxicities, not constituting a safety risk by investigator judgment are allowed.
* Participant has a known additional malignancy that progressed or required active treatment within the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Arms A, B, C, I: Number of Participants with dose-limiting toxicities (DLTs) | Up to 21 days
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 27 months

SECONDARY OUTCOMES:
Number of Participants With Clinically Significant Changes in Laboratory Parameters, Electrocardiogram (ECG) and Vital Signs | Up to 24 months
Number of Participants With Dose Reductions or Delays | Up to 24 months
Number of Participants With Withdrawals due to AEs | Up to 27 months
  Number of participants with adverse events leading to permanent discontinuation of study treatment or withdrawal from study by overall frequency will be assessed.
Overall Response Rate (ORR) | Up to 24 months
  Objective response rate will be calculated as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. It is defined as the percentage of participants with a best overall confirmed complete response (CR) or partial response (PR) at any time as per disease-specific criteria.
Number of Participants With Positive Antidrug Antibodies (ADA) to remzistotug | Up to 27 months
Titres of ADA to remzistotug | Up to 27 months
Number of Participants With Positive ADA to Dostarlimab | Up to 27 months
Titers of ADA to Dostarlimab | Up to 27 months
Number of Participants With Positive ADA to belrestotug | Up to 27 months
Titers of ADA to belrestotug | Up to 27 months
Number of Participants With Positive ADA to nelistotug | Up to 27 months
Titers of ADA to nelistotug | Up to 27 months
Number of Participants With Positive ADA to GSK5764227 | Up to 27 months
Titers of ADA to GSK5764227 | Up to 27 months
Serum Concentrations of remzistotug | Up to 4 months
Serum Concentrations of dostarlimab | Up to 4 months
Serum Concentrations of belrestotug | Up to 4 months
Serum Concentrations of nelistotug | Up to 4 months
Serum Concentrations of GSK5764227 | Up to 4 months
Maximum Observed Plasma Concentration (Cmax) of remzistotug Monotherapy | Up to 27 months
Cmax of remzistotug in Combination With Dostarlimab | Up to 27 months
Cmax of remzistotug in Combination With dostarlimab and belrestotug | Up to 27 months
Cmax following administration of dostarlimab with belrestotug | Up to 27 months
Minimum Observed Plasma Concentration (Cmin) of remzistotug Monotherapy | Up to 27 months
Cmin of remzistotug in Combination With Dostarlimab | Up to 27 months
Cmin of remzistotug in Combination With dostarlimab and belrestotug | Up to 27 months
Cmin following administration of dostarlimab with belrestotug | Up to 27 months
Area Under the Plasma Concentration Curve From Time Zero to Last Time of Quantifiable Concentration (AUC[0-t]) of remzistotug | Up to 27 months
AUC(0-t) of remzistotug in Combination With Dostarlimab | Up to 27 months
AUC(0-t) of remzistotug in Combination With dostarlimab and belrestotug | Up to 27 months
AUC(0-t) following administration of dostarlimab with belrestotug | Up to 27 months
AUC From Time Zero to Infinity (AUC[0-infinity]) of Single Dosing of remzistotug | Up to 27 months
AUC(0-infinity) of Single Dosing of remzistotug in Combination with Dostarlimab | Up to 27 months
AUC(0-infinity) of Single Dosing of remzistotug in Combination With dostarlimab and belrestotug | Up to 27 months
AUC(0-infinity) of Single Dosing of remzistotug following administration of dostarlimab with belrestotug | Up to 27 months
Cmax of dostarlimab in Combination With remzistotug | Up to 27 months
Cmax of dostarlimab in combination with GSK5764227 | Up to 27 months
Cmax of dostarlimab in combination with remzistotug and belrestotug | Up to 27 months
Cmax of dostarlimab in combination with belrestotug | Up to 27 months
Cmax of dostarlimab in combination with belrestotug and remzistotug | Up to 27 months
Cmax of dostarlimab in combination with belrestotug and nelistotug | Up to 27 months
China cohort: Cmax of dostarlimab monotherapy | Up to 18 months
Cmin of dostarlimab in Combination With remzistotug | Up to 27 months
Cmin of dostarlimab in combination with GSK5764227 | Up to 18 months
Cmin of dostarlimab in combination with remzistotug and belrestotug | Up to 27 months
Cmin of dostarlimab in combination with belrestotug | Up to 27 months
Cmin of dostarlimab in combination with belrestotug and remzistotug | Up to 27 months
Cmin of dostarlimab in combination with belrestotug and nelistotug | Up to 27 months
China cohort: Cmin of dostarlimab monotherapy | Up to 18 months
AUC(0-t) of dostarlimab in Combination With remzistotug | Up to 27 months
AUC(0-t) of dostarlimab in combination with GSK5764227 | Up to 18 months
AUC(0-t) of dostarlimab in combination with remzistotug and belrestotug | Up to 27 months
AUC(0-t) of dostarlimab in combination with belrestotug | Up to 27 months
AUC(0-t) of dostarlimab in combination with belrestotug and remzistotug | Up to 27 months
AUC(0-t) of dostarlimab in combination with belrestotug and nelistotug | Up to 27 months
China cohort: AUC(0-t) of dostarlimab monotherapy | Up to 18 months
AUC(0-infinity) of dostarlimab in Combination With remzistotug | Up to 27 months
AUC(0-infinity) of dostarlimab in combination with GSK5764227 | Up to 27 months
AUC(0-infinity) of dostarlimab in combination with remzistotug and belrestotug | Up to 27 months
AUC(0-infinity) of dostarlimab in combination with belrestotug | Up to 27 months
AUC(0-infinity) of dostarlimab in combination with belrestotug and remzistotug | Up to 27 months
AUC(0-infinity) of dostarlimab in combination with belrestotug and nelistotug | Up to 27 months
China cohort: AUC(0-infinity) of dostarlimab monotherapy | Up to 18 months
T1/2 of dostarlimab in Combination With remzistotug | Up to 27 months
T1/2 of dostarlimab in combination with GSK5764227 | Up to 18 months
China cohort: T1/2 of dostarlimab monotherapy | Up to 18 months
Cmax of belrestotug in combination with dostarlimab and belrestotug | Up to 27 months
Cmax of belrestotug in combination with dostarlimab | Up to 27 months
Cmax of belrestotug in combination with dostarlimab and remzistotug | Up to 27 months
Cmax of belrestotug in combination with dostarlimab and nelistotug | Up to 27 months
Cmin of belrestotug in combination with dostarlimab and belrestotug | Up to 27 months
Cmin of belrestotug in combination with dostarlimab | Up to 27 months
Cmin of belrestotug in combination with dostarlimab and remzistotug | Up to 27 months
Cmin of belrestotug in combination with dostarlimab and nelistotug | Up to 27 months
AUC (0-t) of belrestotug in combination with dostarlimab and belrestotug | Up to 27 months
AUC (0-t) of belrestotug in combination with dostarlimab | Up to 27 months
AUC (0-t) of belrestotug in combination with dostarlimab and remzistotug | Up to 27 months
AUC (0-t) of belrestotug in combination with dostarlimab and nelistotug | Up to 27 months
AUC (0-infinity) of belrestotug in combination with dostarlimab and belrestotug | Up to 27 months
AUC (0- infinity) of belrestotug in combination with dostarlimab | Up to 27 months
AUC (0- infinity) of belrestotug in combination with dostarlimab and remzistotug | Up to 27 months
AUC (0- infinity) of belrestotug in combination with dostarlimab and nelistotug | Up to 27 months
Cmax of nelistotug in combination with dostarlimab and belrestotug | Up to 27 months
Cmin of nelistotug in combination with dostarlimab and belrestotug | Up to 27 months
AUC (0-t) of nelistotug in combination with dostarlimab and belrestotug | Up to 27 months
AUC (0-infinity) of nelistotug in combination with dostarlimab and belrestotug | Up to 27 months
Cmax of GSK5764227 in combination with dostarlimab | Up to 18 months
Cmin of GSK5764227 in combination with dostarlimab | Up to 18 months
AUC (0-t) of GSK5764227 conjugated Ab in combination with dostarlimab | Up to 18 months
AUC (0-t) of GSK5764227 small molecule toxin in combination with dostarlimab | Up to 18 months
AUC (0-infinity) of GSK5764227 conjugated Ab in combination with dostarlimab | Up to 18 months
AUC (0-infinity) of GSK5764227 small molecule toxin in combination with dostarlimab | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (7):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- GSK Investigational Site, Nedlands, Western Australia, Australia
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
- China (4):
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuhan
- France (2):
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
- Japan (2):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Seoul, South Korea
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
- United Kingdom (2):
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com